CLINICAL TRIAL: NCT05857436
Title: Relationship of MMP-9 With the Clinical Course of Apical Periodontitis and the Main Bacterial Species in the Oral Microbiota
Brief Title: Relationship Apical Periodontitis and the Main Bacterial Species in the Oral Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seyda Ersahan, DDS, PhD (Other)
Responsible Party: Sponsor-Investigator, Seyda Ersahan, DDS, PhD, Principal Investigator, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Oral Microbiota
Record Dates: First submitted 2023-04-26; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Periapical Periodontitis; MMP-9
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- apical periodontitis (Experimental): 60 patients with AP and extraction indication (due to restorative causes and lesion size) were included in the study
  Interventions: Other: apical periodontitis
- control (Experimental): A total of 30 volunteers who were determined to be systemically and orally healthy (not having AP indication), were included in the study as the control group.
  Interventions: Other: apical periodontitis

INTERVENTIONS:
Other: apical periodontitis — Of these patients, 60 patients with AP and extraction indication (due to restorative causes and lesion size) were included in the study

SUMMARY:
Aim: Apical periodontitis(AP) caused by root canal infection is the most frequent pathological lesion in the jaws. Bacterial products, host immune cells and biologically active factors called locally produced cytokines(such as IL-1, TNF-α) have been reported to play an important role in the pathogenesis of AP. Metalloproteinases(MMP), is a measurable biomarker that plays an important role in the degradation and regeneration of collagen and is an indicator of collagen. This study aimed to determine the main bacterial species in the microbiota as Gr(+) and Gr(-) and to compare the relationship between MMP-9 and TNF-α with controlled patient groups. Methodology:60 patients with AP and extraction indication were included in the study. 30 systemically and orally healthy volunteers were selected as the control group. After access cavity preparation, an initial microbiologic sample(S1) was taken from the root canal. After atraumatic extraction of the tooth, second microbial sample(S2) was taken from the external root surface. After bacterial DNA extraction, 16S rRNA gene primer was designed for sequence analysis. Bacterial community profiling was made by Sanger sequencing of the PCR products. Besides, blood samples were collected from all of the patients. Enzyme-linked immunosorbent assay was used to measure levels of MMP-9 and TNF-α.

DETAILED DESCRIPTION:
60 patients with AP and extraction indication were included in the study. 30 systemically and orally healthy volunteers were selected as the control group. After access cavity preparation, an initial microbiologic sample(S1) was taken from the root canal. After atraumatic extraction of the tooth, second microbial sample(S2) was taken from the external root surface. After bacterial DNA extraction, 16S rRNA gene primer was designed for sequence analysis. Bacterial community profiling was made by Sanger sequencing of the PCR products. Besides, blood samples were collected from all of the patients. Enzyme-linked immunosorbent assay was used to measure levels of MMP-9 and TNF-α Approximately 450 patients who applied to xxxx University, Faculty of Dentistry, Endodontics Department for routine examination due to apical periodontitis complaints were examined and their demographic characteristics were recorded. Patients who had any acute or chronic inflammatory disease, known infection status, history of trauma or surgical operation within 6 months that may affect MMP-9 levels, pregnant and/or lactating, malignity, morbid obesity, arthritis, immunologic diseases, cardiovascular diseases or use of vitamins with high biotin were not included in the study. Additionally, patients who used antibiotics or anti-inflammatory drugs within the last 6 months, and patients with periodontal disease were excluded from the study. Of these patients, 60 patients with AP and extraction indication (due to restorative causes and lesion size) were included in the study. A total of 30 volunteers who were determined to be systemically and orally healthy (not having AP indication), were included in the study as the control group. The study was conducted between March 2022 and February 2023.

Demographic Characteristics & Clinical and Radiographic Evaluation Laboratory Analysis ELISA measurement procedure of MMP-9 and TNF-α levels Bacteriological Sampling from the Root Canal System and Outer Root Surface Genomic DNA Isolation and Measurement of DNA Concentration PCR (16S Universal primer) Purification and sequencing of the 16S rRNA gene Power Analysis and Sample Size Calculations

ELIGIBILITY:
Inclusion Criteria:

* AP and extraction indication (due to restorative causes and lesion size) were included in the study

Exclusion Criteria:

* Patients who had any acute or chronic inflammatory disease, known infection status, history of trauma or surgical operation within 6 months that may affect MMP-9 levels, pregnant and/or lactating, malignity, morbid obesity, arthritis, immunologic diseases, cardiovascular diseases or use of vitamins with high biotin were not included in the study. Additionally, patients who used antibiotics or anti-inflammatory drugs within the last 6 months, and patients with periodontal disease were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Laboratory Analysis | The study was conducted between March 2022 and February 2023
  Blood samples were collected from the patients for MMP-9 and TNF-α analysis. The blood samples taken from the patients in a tube with a gel separator were kept at room temperature for 20-30 minutes to coagulate, and then centrifuged at 1800 g for 10 minutes. T

SECONDARY OUTCOMES:
Bacteriological Sampling from the Root Canal System and Outer Root Surface | The study was conducted between March 2022 and February 2023
  After plaque removal and rubber dam isolation, the operative field was cleaned with 3% hydrogen peroxide and disinfected with 2.5% NaOCl solution. Then, old coronal restorations if present and carious defects were removed, and an access preparation was completed when the root canal space was properly exposed. Afterwards, the tooth (including the pulp chamber), clamp and adjacent rubber dam were once again disinfected with 2.5% NaOCl, followed by inactivation with 10% sodium thiosulfate in order to avoid interference with bacteriological sampling. The working length (WL) was established 1-mm short of the apical foramen with an apex locator (Raypex6; VDW GmbH).
ELISA measurement procedure of MMP-9 and TNF-α levels | The study was conducted between March 2022 and February 2023
  BT lab branded Human Matrix Metalloproteinase 9 and Human Tumor Necrosis Factor-α ELISA Kits (Shangai, China) were used to measure MMP-9 and TNF-α levels. The sensitivity of the kits is 15.12 ng/L and 1.520 pg/mL, respectively, and the measuring range of the kit is 30 - 9000 ng/L and 3 - 900 pg/mL, respectively. The within-run coefficient of variation is < 10%. In the study, measurements were made using BIO-TEK ELx500 ELISA Reader and BIO-TEK ELx50 (USA) washing devices.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Ersahan, Assoc.Prof., Principal Investigator — IstanbulMedipol University
Locations (1):
- Istanbul Medipol University, Faculty of Dentistry, Istanbul, Esenler, Turkey (Türkiye)